CLINICAL TRIAL: NCT06574893
Title: The Effects of Physical Exercise on Simple Inflammatory Markers, Systemic Immune Inflammation Index, and Systemic Immune Response Index in Patients With Schizophrenia
Brief Title: Physical Exercise on Simple Inflammatory Markers, Systemic Immune Inflammation Index, and Systemic Immune Response Index
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dr. Lutfi Kirdar Kartal Training and Research Hospital (Other Government)
Responsible Party: Principal Investigator, İsmail Koç, Assistant Professor, Dr. Lutfi Kirdar Kartal Training and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Keah_2024
Record Dates: First submitted 2024-08-23; First posted 2024-08-28 (Actual); Last update posted 2025-08-19 (Actual); Status verified 2025-03

CONDITIONS: Schizophrenia; Physical Exercise
MeSH Terms: conditions — Schizophrenia; Motor Activity | interventions — Exercise

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- physical exercise group (Experimental): physical exercise
  Interventions: Other: physical exercise
- control group (No Intervention): no intervention

INTERVENTIONS:
Other: physical exercise — physical exercise
  Arms: physical exercise group

SUMMARY:
Mental health is defined as a state of well-being in which a person can realize their talents, cope with the normal stresses of life, and support society by working efficiently and productively. In other words, mental health is a dynamic internal balance that enables individuals to use their diversity of skills in harmony with the universal values of society.

DETAILED DESCRIPTION:
The aim of this study was to investigate the effect of physical exercise on simple inflammation markers, systemic immune inflammation index and systemic inflammation response index in patients with schizophrenia. No other study examining the effect of exercise on these parameters was found in the literature. Therefore, considering the importance of our study, our findings may contribute to the literature and improvement for mental health systems, especially for people with psychotic disorders such as schizophrenia.

ELIGIBILITY:
Inclusion Criteria:

* Individuals diagnosed with schizophrenia by a physician according to DSM-V criteria
* Individuals with schizophrenia who are 18 -55 years

Exclusion Criteria:

* Those who do not consent to participate in the study Patients with a diagnosis other than schizophrenia Pregnancy Patients with chronic metabolic diseases such as diabetes, heart problems and cancer

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 35 (Actual)
Dates: Start 2024-05-04 (Actual); Primary Completion 2024-08-26 (Actual); Study Completion 2025-03-12 (Actual)

PRIMARY OUTCOMES:
sociodemographic characteristics. | 12 weeks
  It will be asked to fill out a structured questionnaire covering their sociodemographic characteristics.
simple inflammatory markers | 12 weeks
  Index Calculation Based on Complete Blood Count

SECONDARY OUTCOMES:
Positive and Negative Syndrome Scale | 12 weeks
  Positive and Negative Syndrome Scale will be used for detecting positive and negative syndromes

CONTACTS AND LOCATIONS:
Locations (1):
- Kartal Dr Lütfi Kırdar Şehir Hastanesi, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No